CLINICAL TRIAL: NCT05960721
Title: Low-dose Rivaroxaban Monotherapy Versus Guideline Determined Medication Therapy After Left Atrial Appendage Occlusion: a Randomized, Open-label, Multicentre, Superiority Trial
Brief Title: Low-dose NOAC Versus GDMT After LAAO
Acronym: RECORD-III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECORD-III
Record Dates: First submitted 2023-06-28; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: Left atrial appendage occlusion; Anti-coagulation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose novel oral anti-coagulation (NOAC)-based anti-thrombotic therapy (Experimental): HAS-BLED<3: Rivaroxaban 15 mg QD for 3 months, followed by Rivaroxaban 10 mg QD indefinitely
  HAS-BLED≥3: Rivaroxaban 10 mg QD for 3 months, followed by Rivaroxaban 2.5 mg bid indefinitely
  Interventions: Drug: Rivaroxaban 15mg; Drug: Rivaroxaban 10mg; Drug: Rivaroxaban 2.5mg
- Guideline determined medication therapy (GDMT) (Active Comparator): HAS-BLED<3: Rivaroxaban 15 mg QD + Aspirin 100mg QD for 3 months, then Aspirin 100mg QD indefinitely
  HAS-BLED≥3: Aspirin 100mg QD + Clopidogrel 75mg QD for 3 months, then Aspirin 100mg QD indefinitely
  Interventions: Drug: Rivaroxaban 15mg; Drug: Aspirin 100mg; Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Rivaroxaban 15mg — QD
Drug: Aspirin 100mg — QD
  Arms: Guideline determined medication therapy (GDMT)
Drug: Clopidogrel 75mg — QD
  Arms: Guideline determined medication therapy (GDMT)
Drug: Rivaroxaban 10mg — QD
  Arms: Low-dose novel oral anti-coagulation (NOAC)-based anti-thrombotic therapy
Drug: Rivaroxaban 2.5mg — B.I.D
  Arms: Low-dose novel oral anti-coagulation (NOAC)-based anti-thrombotic therapy

SUMMARY:
The increased risk of Atrial fibrillation (AF) regarding thromboembolic stroke is predominantly due to the formation and embolization of clots from within the left atrial appendage (LAA). Percutaneous left atrial appendage occlusion (LAAO) is a nonpharmacological strategy for stroke prevention in patients with AF. Data from randomized trials, including PROTECT-AF, PREVAIL, and Prague-17, have suggested that LAAO has comparable efficacy to warfarin or NOACs. Considering these results, LAAO was recommended by the American College of Cardiology (ACC) and European Society of Cardiology (ESC) guidelines as a non-pharmacological stroke prevention strategy for patients with NVAF who have contraindications or are unsuitable for OAC.

The PROTECT-AF and PREVAIL trials stipulated the use of standardized antithrombotic medications which were designed to minimize the risk of stroke, systemic embolism, or device-related thrombosis. This antithrombotic strategy was subsequently endorsed by the guidelines, briefly, patients with LAAO were discharged on warfarin and aspirin for 45 days post-LAAO, if there was no leak or a leak ≤5 mm under transesophageal echocardiography (TEE) at 45-day follow-up, antithrombotic strategies shall switch to dual antiplatelet therapy (DAPT) until 6 months post-LAAO, and then aspirin thereafter.

Although LAAO was recommended by medical societies, previous patient-level meta-analyses have implied that compared with oral anticoagulation, LAAO had significantly more ischemic strokes, suggesting the inability of LAAO to prevent an ischemic stroke from sources beyond LAA. Will a combined strategy of LAAO and OAC further reduce the risk of stroke? The investigators hypothesized that a long-term low dose-Rivaroxaban (10mg daily) post-LAAO might be a potent supplement to the residue risk of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Non-valvular atrial fibrillation (NVAF) patients with successful left atrial appendage occlusion (LAAO)
2. Eligible for guideline-directed anti-thrombotic therapy
3. Able to understand and provide informed consent and comply with all study medications

Exclusion Criteria:

1. Under the age of 18
2. Unable to give informed consent or currently participating in another trial and not yet at its primary endpoint
3. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice)
4. Concurrent medical condition with a life expectancy of less than two years
5. Haemodynamical unstable
6. Known contraindication to medications such as heparin, antiplatelet or anticoagulation drugs, or contrast
7. Peridevice leak > 5mm as assessed immediately after LAAO or any other procedure-related complications
8. Comorbidities other than atrial ﬁbrillation that required long term use of anticoagulation (such as implanted mechanical valve)
9. Percutaneous coronary intervention (PCI) within 1 year.
10. The patient had or is planning to have any cardiac or non-cardiac interventional or surgical procedure within 30 days prior to or 60 days after the WATCHMAN device implant (e.g., PCI, cardioversion, cardiac surgery)
11. Ongoing overt bleeding
12. Previous stroke/TIA within 30 days of enrolment
13. Symptomatic carotid artery disease
14. Severe renal insufficiency (CrCl≤30ml/min/1.73m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4220 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of the composite endpoint of any death, any stroke, systemic embolism, and The Bleeding Academic Research Consortium (BARC)-defined 3 or 5 bleeding events | 24 months post randomization

SECONDARY OUTCOMES:
Rate of the composite endpoint of any death, any stroke, systemic embolism, and BARC defined 3 or 5 bleeding events | 45 days, 6, 12 months (Time-to-event)
Rate of the composite endpoint of any death, any stroke, systemic embolism | 45 days, 6, 12, 24 months (Time-to-event)
Rate of the BARC type 3 or 5 bleeding events | 45 days, 6, 12, 24 months (Time-to-event)
Rate of the composite endpoint of any death, any stroke, systemic embolism, myocardial infarction (MI) | 45 days, 6, 12, 24 months (Time-to-event)
Rate of any death | 45 days, 6, 12, 24 months (Time-to-event)
Rate of any stroke | 45 days, 6, 12, 24 months (Time-to-event)
Rate of systemic embolism | 45 days, 6, 12, 24 months (Time-to-event)
Rate of myocardial infarction (MI) | 45 days, 6, 12, 24 months (Time-to-event)
Rate of BARC type 2, 3 or 5 bleeding events | 45 days, 6, 12, 24 months (Time-to-event)
Rate of BARC type 2 bleeding events | 45 days, 6, 12, 24 months (Time-to-event)
Rate of BARC type 3 bleeding events | 45 days, 6, 12, 24 months (Time-to-event)
Rate of BARC type 5 bleeding events | 45 days, 6, 12, 24 months (Time-to-event)
Rate of GUSTO defined major bleeding and/or minor bleeding | 45 days, 6, 12, 24 months (Time-to-event)
  Global Use of Strategies to Open Occluded Arteries, (GUSTO) defined major bleeding and/or minor bleeding
Rate of TIMI defined major bleeding and/or minor bleeding | 45 days, 6, 12, 24 months (Time-to-event)
  Thrombolysis in Myocardial Infarction (TIMI) defined major bleeding and/or minor bleeding
Rate of ISTH defined major bleeding and/or clinically relevant minor bleeding | 45 days, 6, 12, 24 months (Time-to-event)
  International Society on Thrombosis and Haemostasis (ISTH) defined major bleeding and/or clinically relevant minor bleeding
Rate of patient adherence to allocated medication | 45 days, 6, 12, 24 months (Binary)
  Adherence is defined as the participant who uses the medication strategies in this trial achieving 80% of the time on the therapeutic range
Scores of the National Institutes of Health Stroke Scale (NIHSS) questionnaire | 45 days, 6, 12, 24 months (Continuous)
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
  The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Scores of the Modified Rankin Scale (mRS) | 45 days, 6, 12, 24 months (Continuous)
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials.
Scores of the 5-level EQ-5D version (EQ-5D-5L) questionnaire | 45 days, 6, 12, 24 months (Continuous)
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D., Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No